CLINICAL TRIAL: NCT03566537
Title: Alterations in Quality of Life After Thyroidectomy for Benign Thyroid Disease
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Papavramidis Theodossis, Assistant Professor of surgery, Aristotle University Of Thessaloniki
Other Study IDs: 26181
Record Dates: First submitted 2018-06-11; First posted 2018-06-25 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Benign Thyroid Nodule; Quality of Life
MeSH Terms: interventions — Thyroidectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients who are going to undergo a thyroid surgery due to symptomatic non-toxic multinodular goiter, uncontrolled thyrotoxicosis or suspicious FNA
  Interventions: Procedure: Thyroidectomy
- Controls: Patients with benign thyroid disease, not undergoing thyroidectomy

INTERVENTIONS:
Procedure: Thyroidectomy — Thyroidectomy
  Groups: Cases

SUMMARY:
To detect any changes in Quality of Life in patients with benign thyroid diseases who undergo thyroidectomy compared to patients with benign thyroid diseases and conservative treatment and healthy subjects.

DETAILED DESCRIPTION:
Benign thyroid diseases are a common public health problem. It has been reported that thyroid diseases can affect Quality of Life (QoL), but this is not easy to be assessed. Therefore, a valid instrument is necessary. Such an instrument is Thyroid-related patient-reported outcomes questionnaire (ThyPRO). ThyPRO has been recently translated and validated in Greek language. The questionnaire consists of 85 items grouped in 14 scales concerning goiter, hypothyroidism, hyperthyroidism and eye symptoms, tiredness, cognitive impairment, anxiety, depression, emotional susceptibility, cosmetic complaints and impaired social, and daily and sex life, as well as overall quality of life.

A few studies have demonstrated that various thyroid therapies may improve some aspects of QoL. The aim of the present study is to address the impact of thyroidectomy in QoL in patients with benign thyroid diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is over 18 years old
2. Patient scheduled for a non-emergency operation
3. Patient diagnosed with benign thyroid disease

Exclusion Criteria:

1. Patient is participating in another clinical trial which may affect this study's outcomes
2. Patient with thyroid cancer
3. Previous operation at the thyroid and parathyroid glands or neck irradiation
4. Patient unable to read and write in Greek

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male or female subjects with benign thyroid diseases 18 years of age or older scheduled for thyroidectomy
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Alterations in Quality of Life after thyroidectomy for benign thyroid disease | 2 years
  To detect any changes in Quality of Life in patients with benign thyroid diseases who undergo thyroidectomy compared to patients with benign thyroid diseases and conservative treatment. The Greek, cross-cultural validated, version of ThyPRO questionnaire will be used, as it comprises a reliable and validated instrument to measure thyroid-related quality of life. The 84 questions of ThyPRO are categorized in 13 scales that involve: goiter, hypothyroidism, hyperthyroidism and eyes symptoms, tiredness, cognitive impairment, anxiety, depressivity, emotional susceptibility, cosmetic complaints and impaired social, and daily and sex life. The scales are all scored and the final scores were transformed to a scale from 0 to 100. Lower scores reflect a better thyroid-related quality of life, whereas higher scores reflect a worse quality of life.

SECONDARY OUTCOMES:
Correlation of alterations in Quality of Life after thyroidectomy for benign thyroid disease with secondary characteristics of the patients | 2 years
  Correlation of alterations in Quality of Life after thyroidectomy for benign thyroid disease with secondary characteristics of the patients ( eg age, thyroid autoimmunity, thyroid function, Vitamin D levels)

CONTACTS AND LOCATIONS:
Overall Officials: Theodosios Papavramidis, Asst. Prof., Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Ahepa Hospital, Thessaloniki, Central Macedonia, Greece

IPD SHARING:
Plan to Share IPD: No